CLINICAL TRIAL: NCT01644812
Title: Lifestyle Interventions for Generalized Anxiety Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Jasper Smits, Ph.D., Associate Professor, Southern Methodist University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-001-SMIJ-N
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Aerobic Exercise; Stretching
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Active Comparator): The exercise intervention is a 12-week program involving 150 minutes of moderate intensity exercise (65-69% of participant's age-predicted [220-age] maximum heart rate) each week. Participants will complete one 50-minute supervised treadmill exercise session in the laboratory and 100 minutes of exercise on their own. These exercises may include walking, jogging, biking, or other forms of aerobic exercise. The at-home exercise regimen will be individualized for each participant.
  Interventions: Behavioral: Aerobic exercise
- stretching (Sham Comparator): The exercise intervention is a 12-week program involving 150 minutes of stretching each week (one 50-minute stretching session in the laboratory and 100 minutes of stretching at home). Participants in the stretching condition will work with a facilitator to create a stretching regimen for 100 minutes of home stretching throughout the week. The facilitator will provide a list of potential stretches with descriptions on how to perform them.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic exercise
  Arms: Aerobic exercise
Behavioral: Stretching
  Arms: stretching

SUMMARY:
This two-site (Southern Methodist University (SMU) and Boston University (BU)) study aims to examine the effectiveness of exercise interventions for the treatment of generalized anxiety disorder (GAD). If effective, the use of exercise as a component of treatment for GAD would have a significant public health impact. In addition to improving GAD treatment outcome, exercise is expected to offer health benefits and promote further lifestyle changes.

The present study involves the randomization of 52 adults with GAD to either a 12-week combined supervised- home-based moderate-intensity aerobic exercise protocol (EX) or a 12-week combined supervised- home-based stretching protocol (CTRL). The investigators hypothesize that participants in the EX intervention will evidence greater improvements in anxiety symptoms and quality of life relative to individuals receiving the control intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, ages 18-65.
* Principal diagnosis of Generalized Anxiety Disorder.
* Willing to and capable of providing informed consent, attending all study visits, and complying with the protocol.
* Classified as either being at low risk or moderate risk for cardiovascular disease according to American College of Sports Medicine (ACSM) risk stratification guidelines (see "Telephone Prescreen and Risk Stratification" section for more information).
* Sedentary as defined by ACSM guidelines as not participating in at least 30 minutes of moderate-intensity exercise on at least 3 days a week for at least 3 months.

Exclusion Criteria:

* Currently suicidal or high suicide risk, current or past psychotic disorders of any type, bipolar disorder (I, II, or NOS), schizophrenia or schizoaffective disorder, anorexia, bulimia. Alcohol or drug dependence, abuse of depressants, dissociative anesthetics, hallucinogens, opioids, and cocaine within the last 6 months. Comorbid psychiatric conditions that are relative or absolute contraindications to the use of any treatment option in the protocol.
* Cognitive behavioral therapy within three months of baseline, or ongoing supportive therapy directed specifically toward the treatment of anxiety or mood disorder.
* Psychotropic medications are acceptable only if they are stabilized for at least 3 weeks prior to the baseline visit, as long they are not considered a relative or absolute contraindication to the use of any treatment option in the protocol.
* For women, currently pregnant, plans to be pregnant in the next year, or currently breastfeeding.
* Insufficient command of the English language (i.e., they cannot carry on a conversation with an interviewer in the English language or read associated text).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Penn State worry Questionnaire | changes from baseline to week 13
  The PSWQ is a 16-item inventory designed to capture the generality, excessiveness, and uncontrollability of pathological worry. It has been shown to have good internal consistency with samples consisting of older adults with GAD
GAD-7 | changes from baseline to week 13
  The GAD-7 is a self-reported questionnaire for screening and severity measurement of generalized anxiety disorder (GAD). The researchers conclude that the "GAD-7 is a valid and efficient tool" to screen for anxiety and to assess "its severity in clinical practice and research."
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) | changes from baseline to week 13
  This questionnaire rates 16 aspects of quality of life, including physical health, mood, activities of daily living, and overall life satisfaction. The Q-LES-Q will be used to examine changes in quality of life with treatment.
Clinical Global Impressions Improvement/Severity (CGI) | changes from baseline to week 13
  The CGI-I is a measure of global improvement rated from 1 (very much improved) to 7 (very much worse). The CGI-S measures global severity rated from 1 (not ill) to 7 (extremely ill).

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) | changes from baseline to week 13
  The BAI is a commonly used 21-item, self-report inventory designed to measure severity of anxiety symptoms.
Beck Depression Inventory (BDI) | changes from baseline to week 13
  The BDI is a widely used 21-item, self-report inventory designed to measure severity of depressive symptoms.
Anxiety Sensitivity | changes from baseline to week 13
  Anxiety sensitivity was measured using the Anxiety Sensitivity Index a 16-item questionnaire designed to assess one's tendency to respond fearfully to anxiety-related symptoms. Data on the reliability and validity of the ASI scales have been favorable .
Social Physique Anxiety | changes from baseline to week 13
  The SPAS is a 7-item scale measuring individual anxiety regarding one's figure or physique.

OTHER OUTCOMES:
Health and Risk Assessment Screening. | screening week 0
  The American College of Sports Medicine risk stratification health screening (see Appendix) is a self-guided review of health and medical history for known diseases and signs, symptoms, and risk factors for cardiovascular disease. Female participants will also be administered a pregnancy test.
Psychiatric Diagnoses | Screening week 0
  Diagnostic exclusions and lifetime prevalence of Axis I diagnoses will be determined by the Structured Clinical Interview for DSM-IV non-patient version (SCID-NP; First et al., 2004) during Screening Visit 1. The SCID will be administered during by trained doctoral-level interviewers and will be supervised by the PIs, as has been done successfully in the past (e.g., Zvolensky, Leen-Feldner et al., 2004; Smits et al., 2009).
The Columbia Suicide Severity Rating Scale (C-SSRS) | Screening week 0
  C-SSRS is a standardized measure of current and past self-injurious behavior, suicidal intent, and suicidal behaviors. The C-SSRS has demonstrated good reliability and validity (Hammad et al., 2006; Posner et al., 2007). The C-SSRS will be administered at the Screening Visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - BU Center for Anxiety and Related Disorders, Boston University, Boston, Massachusetts
  - Anxiety Research and Treatment Program, SMU Department of Psychology, Dallas, Texas